CLINICAL TRIAL: NCT04328857
Title: Experimentation of Sensorized Pseudoelastic Orthoses Produced by Additive Manufacturing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: CNR - ICMATE UOS di Lecco (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 686
Record Dates: First submitted 2020-02-27; First posted 2020-03-31 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Upper limb rehabilitation with pseudoelastic orthosis
  Interventions: Device: pseudoelastic orthosis
- Control (No Intervention): Upper limb rehabilitation without pseudoelastic orthosis

INTERVENTIONS:
Device: pseudoelastic orthosis — The subject will be given specific physiotherapy including activities oriented to multimodal exploration and refinement of gross and fine motor skills, customized according to the functional status of the individual patient.
  Arms: Treatment

SUMMARY:
The proposed clinical investigation plan is a pivotal controlled study with two parallel groups, has a total duration of 12 months and involves the recruitment of 34 pediatric patients suffering from acquired brain injury.

The primary objective of the clinical study is to evaluate the improvement of joint stiffness through the use of sensorized pseudoelastic orthoses for the rehabilitation of pediatric patients with acquired brain injury.

The effectiveness of the treatment in terms of joint stiffness (primary outcome) will be assessed and the effect of the treatment will be quantified with clinical evaluation scales and instrumental measurements by means of an optoelectronic system and isokinetic machine. The tolerability and acceptability of the device will also be checked.

ELIGIBILITY:
Inclusion Criteria:

1. Quadriplegia or acquired hemiplegia.
2. Age 6-20 years.
3. Dystonic, dyskinetic, spastic.
4. Chronic phase patients (> 1 year post event).
5. Spastic syndrome with Ashworth Score (AS) for the limb of interest> 1.
6. Collaborative.

Exclusion Criteria:

1. Fixed limitations of the joint.
2. Joint pain.
3. Skin allergies.
4. Behavioral and psychiatric disorders (eg, emotional problems, anxiety, panic attacks).

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Joint Stiffness of affected upper limb joint | After 4 weeks of treatment
  Quantitative measure performed by means of an isokinetic machine (Unit of measure: Nm/°). Changes in joint stiffness following the use of new customized devices during a rehabilitation treatment period. Lower stiffness is better.

SECONDARY OUTCOMES:
Modified Ashworth Scale | After 4 weeks of treatment
  Clinical scale for spasticity (5 levels), higher is worse.
Melbourne Upper Limb Assessment 2 | After 4 weeks of treatment
  Clinical scale for evaluating quality of upper limb movement (16 items, each assessed from 0 to 4 points). Result reported in %. Higher is better.
Quality of Upper Extremity Skills Test | After 4 weeks of treatment
  Clinical scale evaluating the quality of upper extremity function (33 items, 4 domains). Minimum score 0, maximum score 100. Higher is better.
Active range of motion | After 4 weeks of treatment
  Measured with goniometer in degrees.
Passive range of motion | After 4 weeks of treatment
  Measured with goniometer in degrees.
Range of motion of target joint during a pointing-forward task | After 4 weeks of treatment
  Measured in degrees. A kinematic analysis will be performed during a pointing-forward task using an optoelectronic system.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No